CLINICAL TRIAL: NCT00235131
Title: A Clinical Investigation of the Cordis S.M.A.R.T. ™ CONTROL ™ Nitinol Stent System Versus the Bard® Luminexx™ 6F Vascular Stent for the Treatment of TASC C & D Superficial Femoral Artery Long Lesions
Brief Title: The Study to Compare the Cordis SMART™ Stent System With the Bard® Luminexx™ Stent
Acronym: SUPER SL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EE04-02
Record Dates: First submitted 2005-10-04; First posted 2005-10-10 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Arterial Occlusive Diseases
Keywords: Peripheral Artery Occlusive Disease
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cordis S.M.A.R.T.™ CONTROL™ Nitinol Stent System
  Interventions: Device: Smart Stent
- 2 (Active Comparator): Bard® Luminexx™ 6F Vascular Stent
  Interventions: Device: Luminexx Stent

INTERVENTIONS:
Device: Smart Stent — Cordis S.M.A.R.T.™ CONTROL™ Nitinol Stent System
  Arms: 1
Device: Luminexx Stent — Bard® Luminexx™ 6F Vascular Stent
  Arms: 2

SUMMARY:
This study will look at the performance of the Cordis S.M.A.R.T.™ CONTROL ™ Nitinol Stent System for the treatment of TASC C & D superficial femoral artery long lesions (up to 22 cm) in comparison with the Bard® Luminexx™ 6F Vascular Stent as determined by the primary patency rate at 6 and 12 months post procedure.

DETAILED DESCRIPTION:
This is a German multi-center prospective, randomized, two-arm study evaluating performance of the Cordis S.M.A.R.T.™ CONTROL ™ Nitinol Stent System as compared to the C.R. Bard® Luminexx™ 6F Vascular Stent. Patients will be randomized on a 1:1 basis. It is anticipated that a total of 200 patients will be entered into the study.

The study population will consist of approximately 200 symptomatic peripheral vascular disease patients with TASC C & D SFA lesions. The disease will consist of symptomatic, long de novo or restenotic lesions (> 70% stenosis) and occlusions (5 - 22 cm) on diagnostic imaging. The lesion must not extend into the distal SFA and the popliteal artery. At least one distal popliteal artery must be patent as well as one calf vessel. Reference vessel diameter must be >= 4.0 to <= 6.0 mm.

Trial participants will be randomized to the Cordis S.M.A.R.T.™ CONTROL™ Nitinol Stent System or to the Bard® Luminexx™ 6F Vascular Stent.

Patients will be followed for twelve months post-procedure. Study examinations will be done at screening, procedure time, discharge, six, and twelve months post procedure.

This study will be conducted over up to 15 investigational sites in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic leg ischemia by Rutherford classification (category 2, 3, 4 or 5); duration of intermittent claudication (category 2-3) should be at least 3 months.
* One superficial femoral artery de novo or restenotic lesion (more than 70% stenosis or occlusions), with a lesion length of more than 5 to less than 22 cm.
* Patent popliteal artery on the index side, i.e., single vessel runoff or better with at least one of three vessels patent to the lower 1/3 of the calf prior to the day of the procedure.

Exclusion Criteria:

* Revascularisation involving the same limb within 30 days prior to the index procedure or a planned revascularisation within 30 days after the index procedure.
* Patients having total occlusions of the iliac artery on the same side must be excluded.
* Previously implanted stent(s) in the to be treated artery at the same site.
* Requiring stent placement in the distal superficial femoral artery and the popliteal artery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
primary patency detectable by duplex ultrasound through the index lesion | 12 months

SECONDARY OUTCOMES:
technical success | time of deployment
procedural success | up to removal of catheter sheath
procedural complications | up to removal of catheter sheath
Ankle Brachial Index | discharge and 12 months
primary patency | 6 months
binary restenosis | 6 and 12 months
stent fractures | 6 and 12 months
target lesion revascularisation | 6 and 12 months
target vessel revascularisation | 6 and 12 months
adverse events | baseline, discharge, 6 and 12 months post procedure
clinical categorization of chronic limb ischemia by means of the Rutherford classification | discharge, 6 and 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Schneinert, MD, Principal Investigator — Heart Center Leipzig - University Hospital; Stephan Duda, MD, Principal Investigator — Gemeinschaftspraxis füsar Radiologische
Locations (2):
- Germany (2):
  - Gemeinschaftspraxis füsar Radiologische Diagnostik& Zentrum für Minimal Invasite Therapie am Jüdischen Krankenhaus Berlin, Berlin
  - Universitat Leipzig Herzzentrum Abt. Für Klinische u. Intervent. Angiologie, Leipzig